CLINICAL TRIAL: NCT01936597
Title: Prospective Study of 3 Phone Assistance Strategies to Achieve a Continuous Cardiac Massage During Training in Non-hospital Cardiac Cases.
Brief Title: Prospective Study of 3 Phone Assistance Strategies to Achieve a Continuous Cardiac Massage
Acronym: TeleMacc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2012/182/HP; 2012-A01257-36 (Other: ID- RCB number)
Record Dates: First submitted 2013-09-02; First posted 2013-09-06 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Cardiac Arrest
Keywords: external cardiac massage, medical hotline,
MeSH Terms: conditions — Heart Arrest | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single set (control Arm) (Active Comparator): method of external cardiac massage incentive based on a single set. Intervention : Therapeutic and preventive strategies
  Interventions: Other: Therapeutic and preventive strategies
- Controller (Experimental): Audio continuous guidance method by the controller. Intervention : Therapeutic and preventive strategies
  Interventions: Other: Therapeutic and preventive strategies
- Audio (Experimental): Audio continuous guidance method by the controller relayed by an audio. Intervention : Therapeutic and preventive strategies
  Interventions: Other: Therapeutic and preventive strategies

INTERVENTIONS:
Other: Therapeutic and preventive strategies — Single set (control Arm)
  Arms: Single set (control Arm)
Other: Therapeutic and preventive strategies — Controller
  Arms: Controller
Other: Therapeutic and preventive strategies — Audio
  Arms: Audio

SUMMARY:
This study must evaluate the benefit of a continuous audio guidance on the effectiveness of MCE directed by a volunteer.

The evaluation of the MCE for this study is based on both quantitative criteria (based on the recommendations ERC 2010)

* frequency
* depth of chest compressions.

This study compares two methods of continuous audio guide (one arm with an audio continuous guidance method by the regulator and second arm with an audio continuous guidance method by the controller relayed by an audio) to a method of incentive MCE based on a unique set made by the regulator(control arm).

ELIGIBILITY:
Inclusion Criteria:

- Healthy volunteers from the general population understanding the French language.

Exclusion Criteria:

* major physical disability;
* do not speak French
* first aid training under one year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-09; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
frequency and depth of chest compressions | at the end of the simulation (10 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Cédric DAMM, Doctor, Principal Investigator — CHU - Hôpitaux de Rouen
Locations (1):
- CHU - Hôptaux de Rouen (Hôpital Charles Nicolle), Rouen, France